CLINICAL TRIAL: NCT01611038
Title: Chemoprevention of Breast and Prostate Cancers in Shift Workers by Dietary Methylselenocysteine: Effects on Circadian Rhythm and Estrogen Receptor-B Cycling
Brief Title: Methylselenocysteine Effects on Circadian Rhythm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Howard M. Kipen, MD, MPH, Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 0220100243
Record Dates: First submitted 2012-05-18; First posted 2012-06-04 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms | interventions — selenomethylselenocysteine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo given daily
  Interventions: Dietary Supplement: Placebo
- Methylselenocysteine (Experimental): Methylselenocysteine given daily
  Interventions: Dietary Supplement: Methylselenocysteine

INTERVENTIONS:
Dietary Supplement: Methylselenocysteine — Methylselenocysteine capsule given daily
  Arms: Methylselenocysteine
Dietary Supplement: Placebo — Placebo capsule given daily
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine if vitamin supplementation with a naturally occurring dietary amino acid called organic selenium (i.e., methylselenocysteine) can restore disruption of circadian rhythm in shift workers.

DETAILED DESCRIPTION:
All living cells have a circadian (daily) rhythm which controls a variety of bodily functions that change throughout the day, including body temperature, sleep, hunger, activity, hormone levels, etc. The circadian rhythm of the body is controlled by the amount of light that enters our eyes, so on our planet the length of the rhythm is 24 hours long. It is therefore reasonable to suspect that upsetting the timing of the rhythm would lead to changes in body function (as commonly experienced in "jet lag") and that prolonged changes might even lead to alterations in bodily functions and contribute to disease. This suggests that people whose service to the community that requires that they often work at night (nurses, doctors, police, hospital staff, firefighters, airline crews, factory workers, etc), might be at elevated risk of developing diseases. Studies have shown that women who do shift work have an elevated risk of breast cancer, probably as a result of altered hormone levels and cycling. Other studies have shown that vitamin supplementation with a naturally occurring dietary amino acid called organic selenium (i.e., methylselenocysteine) can restore this disrupted rhythm and possibly decrease this disease risk. Thus, the purpose of this study is to investigate whether taking daily selenium (i.e., methylselenocysteine) will restore the disrupted circadian rhythm in shift workers.

ELIGIBILITY:
Inclusion Criteria:

* Permanent night shift schedule

Exclusion Criteria:

* Nutritional supplements that contain selenium
* Pregnant
* Breast feeding
* Heart conditions
* Chronic lung disease
* Cancer therapy (current or past)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Determine if selenium (i.e., methylselenocysteine) supplementation can restore disruption of circadian rhythm and estrogen receptor-B levels in shift workers | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Howard M. Kipen, MD, MPH, Principal Investigator — Rutgers, The State University of New Jersey; Helmut Zarbl, MD, Study Chair — Rutgers, The State University of New Jersey
Locations (1):
- Environmental and Occupational Health Sciences Institute, Piscataway, New Jersey, United States